CLINICAL TRIAL: NCT00647504
Title: Nordic IVUS Study: Prospective Clinical Observational Registry Study Including Consecutive Patients With Clinical Signs or Symptoms Due to In-stent Restenosis (ISR) or Definite (ARC Criteria) Stent Thrombosis (ST)
Brief Title: Prospective Clinical Observational Registry Including Consecutive Patients With In-stent Restenosis or Stent Thrombosis
Acronym: NIVUS
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Saila Vikman, MD,, Tampere University
Other Study IDs: R07054
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Stent Thrombosis; Restenosis
Keywords: stent thrombosis; stent restenosis; intravascular ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Restenosis in Bare metal stent
- 2: Restenosis in Drug eluting stent
- 3: Stent thrombosis
- 4: Control group

SUMMARY:
Prospective clinical observational registry study including consecutive patients with clinical signs or symptoms due to in-stent restenosis (ISR) or definite (ARC criteria) stent thrombosis (ST).

Study hypothesis:

Initial Stent implantation quality (due to technique/problems) are possible major determinants of ST and ISR in real life practice.

Both early, late, and very late ST, and ISR are important factors for long term outcome after initial stent implantation.

Primary objective:

* To elucidate the possible cause(s) of thrombosis or restenosis after stent implantation in real life practice by clinical, angiographic and IVUS evaluation.

Secondary objective:

* To describe the clinical manifestation [stable angina pectoris (AP), unstable AP, non-ST-elevation myocardial infarction (NSTEMI), or ST-elevation MI] of the index event (inclusion).
* To describe the characteristics of patient, lesion and procedure of the initial percutaneous coronary intervention (PCI).
* To describe the antithrombotic pharmacological therapy preceding the index event.
* To describe clinical outcome (death, MI, revascularization, CCS angina class) following treatment of the index event during 12 month follow-up.
* To describe safety of the IVUS procedure (product or procedural related complications/ malfunctions).

DETAILED DESCRIPTION:
Investigational sites:

10-15 high volume Nordic PCI centres with experience in intravascular ultrasound (IVUS).

Patients:

* All consecutive patients admitted with an ischemic event due to ST (estimated number of patients >100) either with BMS or DES.
* All consecutive patients with symptoms or signs of ischemia due to in-stent restenosis with DES (target about 200 patients) and respective BMS patients up to maximum 100 patients.

Total number of patients 400. Control groups 1) Lesions treated during the initial PCI, other than the index lesion, will be used as control lesions for the stent with failure; ST or ISR (IVUS findings).

* The study patients will be compared with a matched population from the Westdenmark Heart Database to compare the patient characteristics and clinical manifestation during initial PCI to find out possible differences in patients with and without stent failure Methods: Detailed description of the characteristics of the patient, lesion and procedure of the index PCI. Thorough description of the antithrombotic pharmacological therapy from index PCI to index event.

Quantitative coronary angiography (QCA) of index lesion at stent implantation and at the index event.

IVUS of the index lesion at the index event.

Logistics A one year workload of 10.000 PCI-patients from 10-15 the participating centres will constitute the population at risk. With a stent thrombosis (definitive stent thrombosis) rate of 1,5 % and a clinical restenosis rate of 4 % there will be 150 patients with any stent thrombosis and 400 patients with any restenosis during a twelve months period. With a DES penetration rate of 50 % about 75 DES-treated patients will experience a stent thrombosis and 200 patients a restenosis.

Ethical approval, data registration and analysis The study will be approved by ethical committees and the data management authorities in the participating Nordic countries.

Data will be registered in a dedicated case report form (CRF).

Continuous variables will be expressed as mean value +SD and discrete variables as absolute values and percentages. Clinical and angiographic variables in the control and index event groups will be compared using the Student's t- and the chi-square tests.

Inclusion criteria Consecutive consented patients with a suspected coronary stent related clinical event, admitted to one of the participating hospitals:

1. Typical symptoms or evidence of myocardial ischemia (stable AP, UAP/NSTEMI, STEMI)
2. Clinical suspicion of ST is based on the ARC criteria (probable ST). ST will be verified by coronary angiography.
3. ISR resulting in clinical symptoms/events (angina pectoris, unstable angina, NSTEMI, STEMI, or documented myocardial ischemia). ISR will be verified by coronary angiography.

IVUS will be performed whenever feasible based on the patient's clinical condition. If IVUS study can not be performed, the above mentioned patients will be included in the initial registry (to evaluate feasibility of IVUS in real life), while final analysis will be based on data obtained from patients with IVUS study performed.

Exclusion criteria:

* Informed consent cannot be obtained. IVUS assessment IVUS will be performed whenever feasible based on the patient's clinical condition primary to treatment of the index lesion. If the IVUS catheter cannot be advanced, the lesion may be dilated by a 2 mm balloon. Mechanical pullback will be used (pull-back speed 0.5 mm/sec). The IVUS examination will be stored on VHS or CD and send to the IVUS core lab. at Odense University Hospital.

All events (technical problems and clinical events) possibly related to the IVUS investigation will be registered and reported following the standard complaint procedure process of the manufacturer. In addition, quarterly progress reports (including complaints) will be provided to the financial supporting company.

QCA The angiography obtained during the index lesion PCI-procedure will be used for qualitative and quantitative coronary angiography (QCA) assessment using a computerized QCA system (Medis, Leiden, Holland).

At the index event angiography, there should be at least two cine-runs before the PCI-procedure and after the procedure with the same angulations as in the index-PCI procedure. The angiograms will be stored on CD and sent to the angiographic core laboratory, Skejby Sygehus, University of Aarhus, Denmark.

End points Primary: Angiographic and IVUS findings:

* procedure related findings at inclusion
* Tabulation and classification of IVUS and angiographic outcomes

Secondary:

* Clinical manifestation of the index event
* IVUS procedure related events Compliance to antithrombotic therapy
* Outcome of treatment (SR and ST) during the 12 month follow-up: clinical status and major cardiac events Safety reporting An appropriate safety plan will be established by the initiating investigator. Relevant procedure, product and study-related events will be reported following the local regulations. Furthermore, any procedural complications and other adverse events as defined by the principle investigator and the study team will be reported to the study coordinator and tracked. The coordinating center and the principle investigator will review tables and listings of all adverse events from the study on a regular basis, analyze these for trends, report unexpected adverse device or procedural events to the appropriate bodies/committees as per local requirements and do an on-going review of the study to ensure patient safety. The coordinating center will follow their procedure for document handling and database reconciliation.

Complaint reporting Device malfunctions, device-related adverse events and product nonconformities will be reported to the appropriate manufacturers following the local product complaint procedures by all participating site(s). Complaints will also be reported to regulatory authorities as per local requirements

ELIGIBILITY:
Inclusion Criteria:

* All Consecutive consented patients with a suspected ST either with BMS or DES. (estimated number of patients >100), admitted to one of the participating hospitals:

  * Typical symptoms or evidence of myocardial ischemia (stable AP, UAP/NSTEMI, STEMI)
  * Clinical suspicion of ST is based on the ARC criteria (probable ST). ST will be verified by coronary angiography.
* All consecutive patients with symptoms or signs of ischemia (angina pectoris, unstable angina, NSTEMI, STEMI, or documented myocardial ischemia) due to ISR with DES (target about 200 patients) and respective BMS patients up to maximum 100 patients.

Exclusion Criteria:

* Informed consent cannot be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10-15 Nordic high volume PCI centers with experience in IVUS.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Tabulation and classification of IVUS outcomes | first day

SECONDARY OUTCOMES:
Clinical manifestation of the index event | 12 months
IVUS procedure related events | 1 week
Outcome of treatment during the 12 month follow-up: clinical status and major cardiac events | 12 months follow-up
Compliance to antithrombotic therapy | 12 month follow-up
Tabulation and classification of angiographic outcomes | first day

CONTACTS AND LOCATIONS:
Overall Officials: Kari Niemelä, MD, CEO, Principal Investigator — Heart Center, Tampere University Hospital
Locations (5):
- Skejby Hospital, Aarhus, Denmark
- Heart Center, Tampere University Hospital, Tampere, Finland
- Riga Heart Center, Riga, Latvia
- Ullevål University Hospital, Oslo, Norway
- Lund University hospital, Lund, Sweden

REFERENCES:
- [Derived] Kosonen P, Vikman S, Jensen LO, Lassen JF, Harnek J, Olivecrona GK, Erglis A, Fossum E, Niemela M, Kervinen K, Ylitalo A, Pietila M, Aaroe J, Kellerth T, Saunamaki K, Thayssen P, Hellsten L, Thuesen L, Niemela K. Intravascular ultrasound assessed incomplete stent apposition and stent fracture in stent thrombosis after bare metal versus drug-eluting stent treatment the Nordic Intravascular Ultrasound Study (NIVUS). Int J Cardiol. 2013 Sep 30;168(2):1010-6. doi: 10.1016/j.ijcard.2012.10.033. Epub 2012 Nov 17. PMID 23164593